CLINICAL TRIAL: NCT03287921
Title: Diagnostic and Therapeutic Approaches to Hyperinflation and Small Airway Disease in COPD
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-hyperinflation
Record Dates: First submitted 2017-09-17; First posted 2017-09-19 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: COPD
Keywords: pulmonary care; COPD; small airway disease; hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- mono bronchodilatation: patients with COPD and features of hyperinflation and small airway disease
  Interventions: Drug: mono bronchodilatation; Drug: dual bronchodilatation
- dual bronchodilatation: patients with COPD and features of hyperinflation and small airway disease
  Interventions: Drug: mono bronchodilatation; Drug: dual bronchodilatation

INTERVENTIONS:
Drug: mono bronchodilatation — within indication according to current GOLD recommendation
  Other Names: bronchodilator monotherapy
Drug: dual bronchodilatation — within indication according to current GOLD recommendation
  Other Names: dual bronchodilator therapy

SUMMARY:
Current guideline-based criteria defining COPD do not meet the challenges set by the complex pathophysiology of the disease. Hyperinflation and affection of the small airways are two components that are not represented in current diagnostic concepts and may relate to early stages of the disease. Moreover, optimal therapeutic interventions in patients with these distinct features remain unclear. The investigators therefore aimed to evaluate novel or not widely used diagnostic approaches for the detection and initiating therapeutic strategies in early stage COPD within the GOLD recommendations.

ELIGIBILITY:
Inclusion Criteria:

* known or first diagnosis of COPD
* lung function testing consistent with hyperinflation or peripheral obstruction
* emphysema in imaging
* symptoms (dyspnea, cough, sputum) and risk factors (>= 10 pack years)
* indication for bronchodilator therapy

Exclusion Criteria:

* GOLD stages 3 and 4 (spirometric)
* indication for dual bronchodilator therapy, triple therapy or inhaled steroid
* contraindication for cardiopulmonary exercise testing
* unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients and out-patients with known or firstly diagnosed COPD
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
residual volume | 8 weeks
  change in residual volume from baseline
D5-20 | 8 weeks
  change in frequency dependence of resistance from baseline
LCI | 8 weeks
  change in lung clearance index from baseline

SECONDARY OUTCOMES:
tpeak | 8 weeks
  increase in exercise duration from baseline
IC | 8 weeks
  increase in inspiratory capacity (isotime and resting) from baseline
SGRQ | 8 weeks
  improvement in St. George's Respiratory Questionaire from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Trinkmann, MD, Principal Investigator — University Medical Center Mannheim
Locations (1):
- University Medical Center Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No